CLINICAL TRIAL: NCT02172092
Title: Fluid Kinetics in Patients With Diabetic Ketoacidosis
Acronym: FDKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Vrinnevi Hospital (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, Associate Professor, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FDKA
Record Dates: First submitted 2014-06-22; First posted 2014-06-24 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Diabetes
Keywords: Diabetes; Ketoacidosis; fluid shift
MeSH Terms: conditions — Diabetes Mellitus; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketoacidosis (Experimental): Patients treated for diabetic ketoacidosis at the Intensive care unit, Vrinnevi Hospital, Norrköping.
  Interventions: Drug: SodiumChloride

INTERVENTIONS:
Drug: SodiumChloride — Infusion of SodiumChloride, blood samples to calculate extracellular volume.

SUMMARY:
The purpose with the study is to follow the fluid shifts that occur during fluid resuscitation of patients with diabetic ketoacidosis.

In the study measurements of changes in blood and urine concentrations of Sodium and Chloride as well as blood hemoglobin are used to mathematically calculate changes in distribution volumes of these different endogenous markers.

DETAILED DESCRIPTION:
Patients treated for diabetic ketoacidosis receive 1000 ml of Sodium Chloride during the first 30 minutes of treatment.

Before, during and after this infusion regular blood samples(and urine) are collected (0, 10, 20, 30, 35, 40, 45, 50, 60, 120, 180 and 300 minutes after infusion start).

B-Hemoglobin, P-Albumine, B-Glucose, P-Sodium, P-Potassium. P-Chlorides, U-Sodium, U-Chloride and U-Glucose. Hourly volume of urine is measured.

The 30 minute infusion can be used to calculate the urine extracellular volume. Thereafter during infusion of Ringers acetate changes in electrolytes in blood as well as urine volume and in the urine excreted electrolytes can be used to calculate the fluid shifts between the different fluid compartments.

Eventually 8 to 12 hours later a second infusion of SodiumChloride is as a control performed.

ELIGIBILITY:
Inclusion Criteria:

* diabetic ketoacidosis needing icu care, conscious patient, signed informed consent.

Exclusion Criteria:

* unconscious patient

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Extracellular volume | 120 minutes
  Masse balance as well as dilution af Sodium and Chloride are used to calculate extracellular volume during an infusion of SodiumChloride. Urine Sodium and Chloride are also measured to register and correct the mass balance.

SECONDARY OUTCOMES:
Distribution of strong and weak acids | 12 hours
  Blood gases are followed. With the Stuart/(Loob) concept it is determined to what degree ketones, lactate or electrolyte shifts influence the acidosis of the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hahn, Prof, Study Director — Linkoeping University
Locations (1):
- Vrinnevi Hospital, Norrköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Svensson R, Hahn RG, Zdolsek JH, Bahlmann H. Plasma volume expansion reveals hidden metabolic acidosis in patients with diabetic ketoacidosis. Intensive Care Med Exp. 2022 Dec;10(1):36. doi: 10.1186/s40635-022-00464-5. Epub 2022 Aug 29. PMID 36038699